CLINICAL TRIAL: NCT01093547
Title: Multi-centre, Open-label, Randomized Trial to Determine the Effect of Icodextrin (Extraneal) Versus Dextrose (Dianeal 2.5%) Used in Long-dwell Exchange, Measuring the HOMA Index in Non-diabetic Prevalent CAPD Patients
Brief Title: Open-label, Randomized Trial to Determine the Effect of Icodextrin Versus Dextrose (Dianeal 2.5%) in HOMA IR
Acronym: ECOS
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Vantive Health LLC (Industry)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ECOS
Record Dates: First submitted 2010-03-24; First posted 2010-03-26 (Estimated); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: End Stage Renal Disease; Continuous Ambulatory Peritoneal Dialysis
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dianeal only (Active Comparator): Patients in Dianeal during the daily exchanges and randomised to Dianeal during the long-dwell exchange
  Interventions: Procedure: Blood samples; Procedure: Measure of peritoneal ultrafiltrates
- Dianeal; Extraneal long-dwell exchange (Active Comparator): Patients in Dianeal during the daily exchanges and randomised to Extraneal during the long-dwell exchange
  Interventions: Procedure: Blood samples; Procedure: Measure of peritoneal ultrafiltrates

INTERVENTIONS:
Procedure: Blood samples — Samples taken monthly
Procedure: Measure of peritoneal ultrafiltrates — Measured by the investigators intermittently and by the patients themselves on a monthly basis

SUMMARY:
Phase IV post-marketing study to evaluate the effect of Extraneal on the HOMA index in non-diabetic CAPD patients over the long-dwell exchange. The purpose of the study is to investigate if the use of Extraneal (which is a mixture of high weight glucose polymers), instead of glucose-based solutions such as Dianeal is going to lower the HOMA index in non-diabetic CAPD patients.

ELIGIBILITY:
Inclusion Criteria:

* must be over 18-years old and under 75-years old
* Peritoneal Equilibration Test (PET) result of high, high average or low average transport
* non-diabetic patient
* be in Continuous Ambulatory Peritoneal Dialysis (CAPD)
* prevalent patients that have been in peritoneal dialysis at least 30 days
* wish to participate

Exclusion Criteria:

* Have a Charlson score of >7 and have a life expectancy of less than 12 months
* HIV positive
* present with peritonitis in the month prior to randomisation
* present with cardiovascular, metabolic or infection complications that have required hospitalisation in the month prior to the randomisation
* have active cancer
* pregnant women
* patients with known allergy to starch-based polymer
* patients who have a significant psychiatric disorder or mental disability that could interfere with the patient´s ability to provide Informed Consent and comply with the protocol procedures
* women incapable of maintaining an effective and accepted contraception method

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-02 (Estimated); Primary Completion 2011-07 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
HOMA index | 4 months
  Measure the changes in the levels of the HOMA index when Extraneal (7.5%) is being administered in the long-dwell exchange and compare these levels to the HOMA index resulting when using Dianeal 2.5% in the long-dwell exchange in non-diabetic CAPD patients. This outcome will be evaluated by measurements taken monthly over a period of 4 months.

SECONDARY OUTCOMES:
HbA1c | 12 months
Ultrafiltration of long-dwell exchange | 12 months
Blood pressure | 12 months
Quality of life | 12 months
Hospitalization rate | 12 months
Time during hospitalization | 12 months
Incidence of Adverse Events | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mauricio R Sanabria, M.D., Principal Investigator — Baxter, RTS Colombia
Locations (1):
- Bogotá, Colombia